CLINICAL TRIAL: NCT06671132
Title: Development and Evaluation of Computerized Chemosensory-Based Orbitofrontal Networks Training for Treatment of Pain (CBOT-Pain) Testing Phase
Brief Title: Development and Evaluation of Computerized Chemosensory-Based Orbitofrontal Networks Training for Treatment of Pain (CBOT-P)
Acronym: CBOT-P-2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Evon Medics LLC (Industry)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Howard University (Other); Global Pain Management, LLC (Unknown); Georgetown University (Other); University of Maryland (Other); Johns Hopkins University (Other); Family and Medical Counseling Service, Inc (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CBOTP2NS125745; 4R44NS125745-02 (NIH)
Record Dates: First submitted 2024-10-28; First posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Chronic Pain; Low Back Pain
Keywords: Chronic pain; Pain; Negative Affect; Cognitive Impairments; Attenuation of Structural Brain Loss in CP with high NA; PACS outcome; Orbitofrontal Cortex; Chemosensory-Based Orbitofrontal Networks Training
MeSH Terms: conditions — Chronic Pain; Low Back Pain; Pain; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- CBOT-P [CBOT + beta caryophyllene (BCP)] (Experimental): CBOT device with BCP
  Interventions: Combination Product: Computerized Chemosensory-Based Orbitofrontal Cortex Training for Pain
- Computerized Chemosensory-Based Orbitofrontal Cortex Training (CBOT) (Sham Comparator): CBOT device
  Interventions: Combination Product: Computerized Chemosensory-Based Orbitofrontal Cortex Training (CBOT)

INTERVENTIONS:
Combination Product: Computerized Chemosensory-Based Orbitofrontal Cortex Training for Pain — CBOT device with beta-caryophyllene
  Other Names: CBOT-P; CBOT device with BCP
  Arms: CBOT-P [CBOT + beta caryophyllene (BCP)]
Combination Product: Computerized Chemosensory-Based Orbitofrontal Cortex Training (CBOT) — CBOT device administering continuous olfactoy stimuli with no BCP
  Other Names: CBOT device
  Arms: Computerized Chemosensory-Based Orbitofrontal Cortex Training (CBOT)

SUMMARY:
The overarching goal of this study phase, Phase II component is to perform a randomized clinical trial of the refined Computerized Chemosensory-Based Orbitofrontal Networks Training for Treatment of Pain [CBOT-Pain (or CBOT-P)] from Phase I, compared to sham Computerized Chemosensory-Based Orbitofrontal Networks Training (CBOT) in Chronic Low Back Pain (CLBP) to determine its short- and long-term effectiveness on Pain, Negative Affect (NA), Cognition and Cortical Brain Structure (PACS), long-term safety, and indications.

The investigators will perform a randomized clinical trial of the refined CBOT-P from Phase I, compared to sham CBOT in CLBP.

Aim 2.1: To determine if CBOT-P significantly influences: (1) acute and long-term reduction of pain severity, and (2) acute and long-term reduction of negative affect. The hypothesis is that optimized CBOT will produce faster, stronger, and longer-lasting improvements in pain severity, NA severity, cognitive impairments, and sleep and functional outcomes.

Aim 2.2 To determine if CBOT-P significantly prevents or reduces progressive shrinkage in the orbitofrontal cortex (OFC), cingulate cortex, and hippocampus. MRI will be acquired at baseline and 6th month. An integrative analysis will be conducted to determine the link between changes in brain structure and cognitive trajectory. The hypothesis is that the CBOT optimized with BCP significantly attenuates shrinkage in OFC and other prefrontal cortex (PFC) regions, compared to the Sham intervention.

DETAILED DESCRIPTION:
The Development and Evaluation of Computerized Chemosensory-Based Orbitofrontal Networks Training for Treatment of Pain (CBOT-P) is a project to develop an effective, scalable, user-friendly, and home-based neuromodulatory platform for broad-spectrum treatment of chronic pain conditions with associated negative affect and cognitive impairments.

The small business, Evon Medics created the olfactory pulsing technology called Computerized Chemosensory-Based Orbitofrontal Cortex Training (CBOT-P) to enable home-based modulation of the OFC and subcortical limbic structures to treat pain and negative affect. In a stakeholder value canvassing exercise chronic pain (CP) sufferers and pain doctors unanimously desire new non-invasive, home-based, safe, and effective interventions that can reduce pain severity by more than 10%, suggesting that current treatments have limitations. Anterograde and retrograde anatomical tracings have been used to demonstrate direct (monosynaptic) anatomical connection between the OFC and the descending inhibitory pain nodes at the midbrain periaqueductal gray matter (PAG). Transition to CP is marked by weakened modulation of the PAG descending inhibition.

In this study phase, Phase II of this Fast-Track SBIR application, the investigators will conduct a multi-site study of 220 adult patients with CLBP to establish stronger evidence that the product controls pain, reduces negative mood, improves cognition, and protects the brain from shrinking in six months of treatment. Participants in this phase will be randomly assigned in a 1:1 ratio to daily treatment with CBOT-P device (i.e., CBOT with beta-caryophyllene (BCP) compared to a control (Sham) device that looks like the device but does not have the active ingredients and the programmed parameters on the ability to improve pain, mood, cognition and brain functions in chronic pain. Structural magnetic resonance imaging (MRI) will be acquired at baseline and after 6 months of daily treatment with optimized CBOT (based on Phase I) or Sham CBOT device to improve masking. Pain and NA measures, Cognitive batteries, and physical and functional measures will be assessed at baseline, months 1, 3, and 6. Participants would be encouraged through mobile health prompts to complete subjective pain, affect, sleep, and functional studies at the end of each study week. CLBP volunteers, radiologists, and clinicians assessing outcome measures will be blinded to these assignments.

The investigators will also collect user experiences to help refine a final marketable CBOT product, enter the FDA breakthrough designation program for pain that would lead to Medicare/Medicaid reimbursement, engage a wider network of pain stakeholders, and establish marketing for commercial success.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18-85.
2. Pain duration > 6 months.
3. Must meet the minimum criteria for cognitive function using the PROMIS 4-item cognitive screener >3.
4. Average pain score of > 5/10, with low back pain being the primary pain site. (5) CLBP (chronic low back pain) meeting Quebec Task Force Classification System Categories I-III.

(6) Evidence of a prior lumbar spine X-ray to rule out red flags, such as infection, tumor, or fracture.

(7) For those taking opioids (the opioid subgroup), participants must be prescribed opioids currently for at least 3 consecutive months prior to enrollment. Such patients must be on opioids for a minimum of three months, taking them daily or intermittently during the week. (8) Subject must agree that opioids cannot be increased during the study. (9) No substance use disorder (SUD), except tobacco in the past year based on substance screening survey and frequent urine toxicology screens. (10) No acute suicidality, mania, or psychosis. This will be assessed at study entry, which will also include a review of history in the EHR, Diagnostic Interview for Genetic Studies (DIGS) and Columbia Suicide Severity Rating scale (C-SSRS) and (11) Finally, participants must sign IRB-approved consent.

Exclusion Criteria:

1. Back surgery within the past six months.
2. Active worker's compensation or litigation claims.
3. New pain and/or psychiatric treatments within 2 weeks of enrollment.
4. Intent to add new or increase pain treatments during the study period, such as back surgery, nerve block procedures, or medications.
5. Intent to add new psychiatric treatments during the first 3 months of the study.
6. Any clinically unstable systemic illness that is judged to interfere with the trial.
7. History of cardiac, nervous system, or respiratory disease that, in the investigator's judgment, precludes participation in the study because of a heightened potential for respiratory depression.
8. Non-ambulatory status.
9. Pregnancy or the intent to become pregnant during the study. Women of childbearing age will have urine pregnancy testing at enrollment and monthly. (10) Anosmia or significant nasal disease

(11) Contraindications to MRI (12) Stroke or TBI (traumatic brain injury).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2024-10-23 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Patient Reported Outcomes Measurement Information System (PROMIS) Numeric Rating Scale v1.0 - Pain Intensity (Aim 2.1) | Baseline to month 1 visit
  Change in 11-point score PROMIS Numeric Rating Scale v1.0 - Pain Intensity from baseline.
  The Numeric Rating Scale measures each consist of a single item rating pain on average over the past 7 days from 0 (no pain) to 10 (worst pain).
Positive and Negative Affect Schedule (PANAS) rating scale (Aim 2.1) | Baseline to month 1 visit
  Change in negative affect score from the PANAS rating scale
  It consists of two 10-item scales to measure both positive and negative affect. Each item is rated on a 5-point scale of 1 (not at all) to 5 (very much).
  Positive Affect Scores can range from 10 - 50, with higher scores representing higher levels of positive affect.
  Negative Affect Scores can range from 10 - 50, with lower scores representing lower levels of negative affect.
Patient Reported Outcomes Measurement Information System (PROMIS) Numeric Rating Scale v1.0 - Pain Intensity (Aim 2.1) | Baseline to month 3 visit
  Change in 11-point score PROMIS Numeric Rating Scale v1.0 - Pain Intensity from baseline.
  The Numeric Rating Scale measures each consist of a single item rating pain on average over the past 7 days from 0 (no pain) to 10 (worst pain).
Positive and Negative Affect Schedule (PANAS) rating scale (Aim 2.1) | Baseline to month 3 visit
  Change in negative affect score from the PANAS rating scale
  It consists of two 10-item scales to measure both positive and negative affect. Each item is rated on a 5-point scale of 1 (not at all) to 5 (very much).
  Positive Affect Scores can range from 10 - 50, with higher scores representing higher levels of positive affect.
  Negative Affect Scores can range from 10 - 50, with lower scores representing lower levels of negative affect.
Patient Reported Outcomes Measurement Information System (PROMIS) Numeric Rating Scale v1.0 - Pain Intensity (Aim 2.1) | Baseline to month 6 visit
  Change in 11-point score PROMIS Numeric Rating Scale v1.0 - Pain Intensity from baseline.
  The Numeric Rating Scale measures each consist of a single item rating pain on average over the past 7 days from 0 (no pain) to 10 (worst pain).
Positive and Negative Affect Schedule (PANAS) rating scale (Aim 2.1) | Baseline to month 6 visit
  Change in negative affect score from the PANAS rating scale
  It consists of two 10-item scales to measure both positive and negative affect. Each item is rated on a 5-point scale of 1 (not at all) to 5 (very much).
  Positive Affect Scores can range from 10 - 50, with higher scores representing higher levels of positive affect.
  Negative Affect Scores can range from 10 - 50, with lower scores representing lower levels of negative affect.
Grey Matter Volumes of OrbitoFrontal Cortex and Hippocampus Aim 2.2 | Baseline and 6 months
  Change in the structural brain MRI baseline grey matter volumes of the orbitofrontal cortex and hippocampus at 6 months.
  The investigators will use linear mixed effect and coefficient measures, and include sex, age, opioid medications, and duration of CP as confounders and as effect modifiers. Investigators will also estimate linear and non-linear trajectories.

SECONDARY OUTCOMES:
Patient Reported Outcomes Measurement Information System (PROMIS) Short Form v1.1 - Pain Interference scores. Aim 2.1 | Baseline to month 1 visit
  Change in PROMIS Short Form v1.1 - Pain Interference scores.
  The PROMIS Pain Interference Short Form 4a is consists of 4 questions, each question usually has five response options ranging in value from one to five. The lowest possible raw score is 4; the highest possible raw score is 20.
  PROMIS instruments are scored using item-level calibrations. Scoring method uses responses to each item for each participant, referred to as "response pattern scoring." Tables showing score conversion are available in the PROMIS manual. Use the applicable table to translate the total raw score into a T-score for each participant. The T-score rescales the raw score into a standardized T-score with a mean of 50 and a standard deviation (SD) of 10. A higher PROMIS T-score represents more of the concept being measured.
Patient Reported Outcomes Measurement Information System (PROMIS) Short Form v1.0 - Anxiety scores Aim 2.1 | Baseline to month 1 visit
  Change in PROMIS Short Form v1.0 - Anxiety scores
  The PROMIS Anxiety 1a is consists of 55 questions, each question usually has five response options ranging in value from one to five. The lowest possible raw score is 55; the highest possible raw score is 275.
  PROMIS instruments are scored using item-level calibrations. Scoring method uses responses to each item for each participant, referred to as "response pattern scoring." Tables showing score conversion are available in the PROMIS manual. Use the applicable table to translate the total raw score into a T-score for each participant. The T-score rescales the raw score into a standardized T-score with a mean of 50 and a standard deviation (SD) of 10. A higher PROMIS T-score represents more of the concept being measured.
Patient Reported Outcomes Measurement Information System (PROMIS) Short Form v1.0 - Sleep Disturbance scores Aim 2.1 | Baseline to month 1 visit
  Change in PROMIS Short Form v1.0 - Sleep Disturbance scores
  The PROMIS Sleep Disturbance v1.0 is consists of 26 questions, each question usually has five response options ranging in value from one to five. The lowest possible raw score is 26; the highest possible raw score is 130.
  PROMIS instruments are scored using item-level calibrations. Scoring method uses responses to each item for each participant, referred to as "response pattern scoring." Tables showing score conversion are available in the PROMIS manual. Use the applicable table to translate the total raw score into a T-score for each participant. The T-score rescales the raw score into a standardized T-score with a mean of 50 and a standard deviation (SD) of 10. A higher PROMIS T-score represents more of the concept being measured.
Total Sleep Time (TST) Centrepoint Insight Actigraph watch Sleep Parameters Aim 2.1 | Baseline and 1 month
  Change in Total Sleep Time (TST) captured by Centrepoint Insight Actigraph watch:
  The total sleep time is the total amount of sleep time scored during the total recording time. This includes time from sleep onset to sleep offset and is distributed throughout the sleep time as minutes of Stage N1 sleep, Stage N2 sleep, Stage N3, and rapid eye movement (REM) sleep. All these times are described in minutes.
  A low total sleep time may indicate that the patient slept for an insufficient period of time due to non-medical/non-physiological reasons, certain medical or sleep disorders, or as a result of the effect of medications. Long total sleep time may suggest prior sleep deprivation, medical conditions, or effects of medications.
Sleep Onset Latency (SOL) Centrepoint Insight Actigraph watch Sleep Parameters Aim 2.1 | Baseline and 1 month
  Change in Sleep Onset Latency (SOL) captured by Centrepoint Insight Actigraph watch:
  Sleep latency is the time in minutes from 'lights out' that marks the starting of total recording time to the first epoch scored as sleep.
  Sleep latency also indicates if reasonable attention was paid to the patient's sleep diary and the 'lights out' time was close to the patient's routine bedtime at home. Clearly, if the lights are turned out earlier than the patient's usual bedtime, sleep latency would be spuriously long, and the patient may not fall asleep until his/her usual sleep time is reached. Similarly, if the 'lights out' time is later than the patient's usual bedtime, the patient will be sleepy and a spuriously short sleep latency will be recorded. It is of utmost importance that the patient's usual habitual sleep time is incorporated into the patient's sleep study design and 'lights out' time is approximated.
Sleep Efficiency (SE) Centrepoint Insight Actigraph watch Sleep Parameters Aim 2.1 | Baseline and 1 month
  Change in Sleep Efficiency (SE) captured by Centrepoint Insight Actigraph watch:
  Sleep efficiency refers to percentage of total time in bed actually spent in sleep calculated as sum of Stage N1, Stage N2, Stage N3, and REM sleep, divided by the total time in bed and multiplied by 100.
  Sleep efficiency gives an overall sense of how well the patient slept, but it does not distinguish frequent, brief episodes of wakefulness. A low sleep efficiency percentage could result from long sleep latency and long sleep offset to lights on time with otherwise normal quantity and quality of sleep in between. Many laboratories report total wake time, that is, the amount of wake time during the total recording time in minutes after the sleep onset. The total amount gives a general estimation for overall quality of sleep. Total wake time is the reciprocal of total sleep time. A high total sleep time percent is always associated with low total wake time percent and vice versa
Wake After Sleep Onset (WASO) Centrepoint Insight Actigraph watch Sleep Parameters Aim 2.1 | Baseline and 1 month
  Change in Wake After Sleep Onset (WASO) captured by Centrepoint Insight Actigraph watch:
  Wake after sleep onset, also known as 'WASO' refers to periods of wakefulness occurring after defined sleep onset. This parameter measures wakefulness, excluding the wakefulness occurring before sleep onset. WASO time is a better reflection of sleep fragmentation.
Patient Reported Outcomes Measurement Information System (PROMIS) Short Form v2.0 - Physical Function Aim 2.1 | Baseline to month 1 visit
  Change in PROMIS Short Form v2.0 - Physical Function score
  PROMIS Physical Function instruments measure self-reported capability rather than actual performance of physical activities. The PROMIS short form v2.0 Physical function instrument is consists of 22 questions, each question has five response options ranging in value from one to five. The lowest possible raw score is 22 and the highest possible raw score is 113.
  PROMIS instruments are scored using item-level calibrations. Scoring method uses responses to each item for each participant, referred to as "response pattern scoring." Tables showing score conversion are available in the PROMIS manual. Use the applicable table to translate the total raw score into a T-score for each participant. The T-score rescales the raw score into a standardized T-score with a mean of 50 and a standard deviation (SD) of 10. A higher PROMIS T-score represents more of the concept being measured.
Patient Global Impression of Change Aim 2.1 | Baseline to month 1 visit
  Change in Patient Global Impression of Change score
  The Patient Global Impression of Change scale is a single, self-administered question asking respondents to rate how their condition has changed since a certain point in time. It is a patient-reported outcome measure that can be used to assess treatment benefit in clinical trials or practice. It is based on the Clinical Global Impression of Change scale, which is an observer-rated scale of symptom severity and treatment response. The scale ranges from 1 (no change or worse) to 7 (a great deal better).
California Verbal Learning Test (CVLT) Aim 2.1 | Baseline to month 1 visit
  The California Verbal Learning Test - Third Edition (CVLT-III) is a comprehensive assessment of verbal learning and memory. It produces a variety of scores, including:
  d' score A raw score that reflects the difference between the hit rate (signal) and the false positive (FP) rate (noise). The d' score is calculated by subtracting the FP rate from the hit rate, after applying a z-transform to each.
  Total RD A score that can range from +4.0 to -4.0. A high score indicates a high number of hits and a low number of FP errors, while a low score indicates a low number of hits and a high number of FP errors.
  Scaled scores Scores that are adjusted for age and gender using the CVLT-3 standardization sample norms.
  T-scores Scores that are derived from scaled scores and demographic information using look-up tables. T-scores are a comparison of an individual's memory performance to what is expected based on their demographics.
Patient Reported Outcomes Measurement Information System (PROMIS) Short Form v1.1 - Pain Interference scores. Aim 2.1 | Baseline to month 3 visit
  Change in PROMIS Short Form v1.1 - Pain Interference scores.
  The PROMIS Pain Interference Short Form 4a is consists of 4 questions, each question usually has five response options ranging in value from one to five. The lowest possible raw score is 4; the highest possible raw score is 20.
  PROMIS instruments are scored using item-level calibrations. Scoring method uses responses to each item for each participant, referred to as "response pattern scoring." Tables showing score conversion are available in the PROMIS manual. Use the applicable table to translate the total raw score into a T-score for each participant. The T-score rescales the raw score into a standardized T-score with a mean of 50 and a standard deviation (SD) of 10. A higher PROMIS T-score represents more of the concept being measured.
Patient Reported Outcomes Measurement Information System (PROMIS) Short Form v1.0 - Anxiety scores Aim 2.1 | Baseline to month 3 visit
  Change in PROMIS Short Form v1.0 - Anxiety scores
  The PROMIS Anxiety 1a is consists of 55 questions, each question usually has five response options ranging in value from one to five. The lowest possible raw score is 55; the highest possible raw score is 275.
  PROMIS instruments are scored using item-level calibrations. Scoring method uses responses to each item for each participant, referred to as "response pattern scoring." Tables showing score conversion are available in the PROMIS manual. Use the applicable table to translate the total raw score into a T-score for each participant. The T-score rescales the raw score into a standardized T-score with a mean of 50 and a standard deviation (SD) of 10. A higher PROMIS T-score represents more of the concept being measured.
Patient Reported Outcomes Measurement Information System (PROMIS) Short Form v1.0 - Sleep Disturbance scores Aim 2.1 | Baseline to month 3 visit
  Change in PROMIS Short Form v1.0 - Sleep Disturbance scores
  The PROMIS Sleep Disturbance v1.0 is consists of 26 questions, each question usually has five response options ranging in value from one to five. The lowest possible raw score is 26; the highest possible raw score is 130.
  PROMIS instruments are scored using item-level calibrations. Scoring method uses responses to each item for each participant, referred to as "response pattern scoring." Tables showing score conversion are available in the PROMIS manual. Use the applicable table to translate the total raw score into a T-score for each participant. The T-score rescales the raw score into a standardized T-score with a mean of 50 and a standard deviation (SD) of 10. A higher PROMIS T-score represents more of the concept being measured.
Total Sleep Time (TST) Centrepoint Insight Actigraph watch Sleep Parameters Aim 2.1 | Baseline and month 3
  Change in Total Sleep Time (TST) captured by Centrepoint Insight Actigraph watch:
  The total sleep time is the total amount of sleep time scored during the total recording time. This includes time from sleep onset to sleep offset and is distributed throughout the sleep time as minutes of Stage N1 sleep, Stage N2 sleep, Stage N3, and rapid eye movement (REM) sleep. All these times are described in minutes.
  A low total sleep time may indicate that the patient slept for an insufficient period of time due to non-medical/non-physiological reasons, certain medical or sleep disorders, or as a result of the effect of medications. Long total sleep time may suggest prior sleep deprivation, medical conditions, or effects of medications.
Sleep Onset Latency (SOL) Centrepoint Insight Actigraph watch Sleep Parameters Aim 2.1 | Baseline and month 3
  Change in Sleep Onset Latency (SOL) captured by Centrepoint Insight Actigraph watch:
  Sleep latency is the time in minutes from 'lights out' that marks the starting of total recording time to the first epoch scored as sleep.
  Sleep latency also indicates if reasonable attention was paid to the patient's sleep diary and the 'lights out' time was close to the patient's routine bedtime at home. Clearly, if the lights are turned out earlier than the patient's usual bedtime, sleep latency would be spuriously long, and the patient may not fall asleep until his/her usual sleep time is reached. Similarly, if the 'lights out' time is later than the patient's usual bedtime, the patient will be sleepy and a spuriously short sleep latency will be recorded. It is of utmost importance that the patient's usual habitual sleep time is incorporated into the patient's sleep study design and 'lights out' time is approximated.
Sleep Efficiency (SE) Centrepoint Insight Actigraph watch Sleep Parameters Aim 2.1 | Baseline and month 3
  Change in Sleep Efficiency (SE) captured by Centrepoint Insight Actigraph watch:
  Sleep efficiency refers to percentage of total time in bed actually spent in sleep calculated as sum of Stage N1, Stage N2, Stage N3, and REM sleep, divided by the total time in bed and multiplied by 100.
  Sleep efficiency gives an overall sense of how well the patient slept, but it does not distinguish frequent, brief episodes of wakefulness. A low sleep efficiency percentage could result from long sleep latency and long sleep offset to lights on time with otherwise normal quantity and quality of sleep in between. Many laboratories report total wake time, that is, the amount of wake time during the total recording time in minutes after the sleep onset. The total amount gives a general estimation for overall quality of sleep. Total wake time is the reciprocal of total sleep time. A high total sleep time percent is always associated with low total wake time percent and vice versa
Wake After Sleep Onset (WASO) Centrepoint Insight Actigraph watch Sleep Parameters Aim 2.1 | Baseline and month 3
  Change in Wake After Sleep Onset (WASO) captured by Centrepoint Insight Actigraph watch:
  Wake after sleep onset, also known as 'WASO' refers to periods of wakefulness occurring after defined sleep onset. This parameter measures wakefulness, excluding the wakefulness occurring before sleep onset. WASO time is a better reflection of sleep fragmentation.
Patient Reported Outcomes Measurement Information System (PROMIS) Short Form v2.0 - Physical Function Aim 2.1 | Baseline to month 3 visit
  Change in PROMIS Short Form v2.0 - Physical Function score
  PROMIS Physical Function instruments measure self-reported capability rather than actual performance of physical activities. The PROMIS short form v2.0 Physical function instrument is consists of 22 questions, each question has five response options ranging in value from one to five. The lowest possible raw score is 22 and the highest possible raw score is 113.
  PROMIS instruments are scored using item-level calibrations. Scoring method uses responses to each item for each participant, referred to as "response pattern scoring." Tables showing score conversion are available in the PROMIS manual. Use the applicable table to translate the total raw score into a T-score for each participant. The T-score rescales the raw score into a standardized T-score with a mean of 50 and a standard deviation (SD) of 10. A higher PROMIS T-score represents more of the concept being measured.
Patient Global Impression of Change Aim 2.1 | Baseline to month 3 visit
  Change in Patient Global Impression of Change score
  The Patient Global Impression of Change scale is a single, self-administered question asking respondents to rate how their condition has changed since a certain point in time. It is a patient-reported outcome measure that can be used to assess treatment benefit in clinical trials or practice. It is based on the Clinical Global Impression of Change scale, which is an observer-rated scale of symptom severity and treatment response. The scale ranges from 1 (no change or worse) to 7 (a great deal better).
California Verbal Learning Test (CVLT) Aim 2.1 | Baseline to month 3 visit
  The California Verbal Learning Test - Third Edition (CVLT-III) is a comprehensive assessment of verbal learning and memory. It produces a variety of scores, including:
  d' score A raw score that reflects the difference between the hit rate (signal) and the false positive (FP) rate (noise). The d' score is calculated by subtracting the FP rate from the hit rate, after applying a z-transform to each.
  Total RD A score that can range from +4.0 to -4.0. A high score indicates a high number of hits and a low number of FP errors, while a low score indicates a low number of hits and a high number of FP errors.
  Scaled scores Scores that are adjusted for age and gender using the CVLT-3 standardization sample norms.
  T-scores Scores that are derived from scaled scores and demographic information using look-up tables. T-scores are a comparison of an individual's memory performance to what is expected based on their demographics.
Patient Reported Outcomes Measurement Information System (PROMIS) Short Form v1.1 - Pain Interference scores. Aim 2.1 | Baseline to month 6 visit
  Change in PROMIS Short Form v1.1 - Pain Interference scores.
  The PROMIS Pain Interference Short Form 4a is consists of 4 questions, each question usually has five response options ranging in value from one to five. The lowest possible raw score is 4; the highest possible raw score is 20.
  PROMIS instruments are scored using item-level calibrations. Scoring method uses responses to each item for each participant, referred to as "response pattern scoring." Tables showing score conversion are available in the PROMIS manual. Use the applicable table to translate the total raw score into a T-score for each participant. The T-score rescales the raw score into a standardized T-score with a mean of 50 and a standard deviation (SD) of 10. A higher PROMIS T-score represents more of the concept being measured.
Patient Reported Outcomes Measurement Information System (PROMIS) Short Form v1.0 - Anxiety scores Aim 2.1 | Baseline to month 6 visit
  Change in PROMIS Short Form v1.0 - Anxiety scores
  The PROMIS Anxiety 1a is consists of 55 questions, each question usually has five response options ranging in value from one to five. The lowest possible raw score is 55; the highest possible raw score is 275.
  PROMIS instruments are scored using item-level calibrations. Scoring method uses responses to each item for each participant, referred to as "response pattern scoring." Tables showing score conversion are available in the PROMIS manual. Use the applicable table to translate the total raw score into a T-score for each participant. The T-score rescales the raw score into a standardized T-score with a mean of 50 and a standard deviation (SD) of 10. A higher PROMIS T-score represents more of the concept being measured.
Patient Reported Outcomes Measurement Information System (PROMIS) Short Form v1.0 - Sleep Disturbance scores Aim 2.1 | Baseline to month 6 visit
  Change in PROMIS Short Form v1.0 - Sleep Disturbance scores
  The PROMIS Sleep Disturbance v1.0 is consists of 26 questions, each question usually has five response options ranging in value from one to five. The lowest possible raw score is 26; the highest possible raw score is 130.
  PROMIS instruments are scored using item-level calibrations. Scoring method uses responses to each item for each participant, referred to as "response pattern scoring." Tables showing score conversion are available in the PROMIS manual. Use the applicable table to translate the total raw score into a T-score for each participant. The T-score rescales the raw score into a standardized T-score with a mean of 50 and a standard deviation (SD) of 10. A higher PROMIS T-score represents more of the concept being measured.
Total Sleep Time (TST) Centrepoint Insight Actigraph watch Sleep Parameters Aim 2.1 | Baseline and month 6
  Change in Total Sleep Time (TST) captured by Centrepoint Insight Actigraph watch:
  The total sleep time is the total amount of sleep time scored during the total recording time. This includes time from sleep onset to sleep offset and is distributed throughout the sleep time as minutes of Stage N1 sleep, Stage N2 sleep, Stage N3, and rapid eye movement (REM) sleep. All these times are described in minutes.
  A low total sleep time may indicate that the patient slept for an insufficient period of time due to non-medical/non-physiological reasons, certain medical or sleep disorders, or as a result of the effect of medications. Long total sleep time may suggest prior sleep deprivation, medical conditions, or effects of medications.
Sleep Onset Latency (SOL) Centrepoint Insight Actigraph watch Sleep Parameters Aim 2.1 | Baseline and month 6
  Change in Sleep Onset Latency (SOL) captured by Centrepoint Insight Actigraph watch:
  Sleep latency is the time in minutes from 'lights out' that marks the starting of total recording time to the first epoch scored as sleep.
  Sleep latency also indicates if reasonable attention was paid to the patient's sleep diary and the 'lights out' time was close to the patient's routine bedtime at home. Clearly, if the lights are turned out earlier than the patient's usual bedtime, sleep latency would be spuriously long, and the patient may not fall asleep until his/her usual sleep time is reached. Similarly, if the 'lights out' time is later than the patient's usual bedtime, the patient will be sleepy and a spuriously short sleep latency will be recorded. It is of utmost importance that the patient's usual habitual sleep time is incorporated into the patient's sleep study design and 'lights out' time is approximated.
Sleep Efficiency (SE) Centrepoint Insight Actigraph watch Sleep Parameters Aim 2.1 | Baseline and month 6
  Change in Sleep Efficiency (SE) captured by Centrepoint Insight Actigraph watch:
  Sleep efficiency refers to percentage of total time in bed actually spent in sleep calculated as sum of Stage N1, Stage N2, Stage N3, and REM sleep, divided by the total time in bed and multiplied by 100.
  Sleep efficiency gives an overall sense of how well the patient slept, but it does not distinguish frequent, brief episodes of wakefulness. A low sleep efficiency percentage could result from long sleep latency and long sleep offset to lights on time with otherwise normal quantity and quality of sleep in between. Many laboratories report total wake time, that is, the amount of wake time during the total recording time in minutes after the sleep onset. The total amount gives a general estimation for overall quality of sleep. Total wake time is the reciprocal of total sleep time. A high total sleep time percent is always associated with low total wake time percent and vice versa
Wake After Sleep Onset (WASO) Centrepoint Insight Actigraph watch Sleep Parameters Aim 2.1 | Baseline and month 6
  Change in Wake After Sleep Onset (WASO) captured by Centrepoint Insight Actigraph watch:
  Wake after sleep onset, also known as 'WASO' refers to periods of wakefulness occurring after defined sleep onset. This parameter measures wakefulness, excluding the wakefulness occurring before sleep onset. WASO time is a better reflection of sleep fragmentation.
Patient Reported Outcomes Measurement Information System (PROMIS) Short Form v2.0 - Physical Function Aim 2.1 | Baseline to month 6 visit
  Change in PROMIS Short Form v2.0 - Physical Function score
  PROMIS Physical Function instruments measure self-reported capability rather than actual performance of physical activities. The PROMIS short form v2.0 Physical function instrument is consists of 22 questions, each question has five response options ranging in value from one to five. The lowest possible raw score is 22 and the highest possible raw score is 113.
  PROMIS instruments are scored using item-level calibrations. Scoring method uses responses to each item for each participant, referred to as "response pattern scoring." Tables showing score conversion are available in the PROMIS manual. Use the applicable table to translate the total raw score into a T-score for each participant. The T-score rescales the raw score into a standardized T-score with a mean of 50 and a standard deviation (SD) of 10. A higher PROMIS T-score represents more of the concept being measured.
Patient Global Impression of Change Aim 2.1 | Baseline to month 6 visit
  Change in Patient Global Impression of Change score
  The Patient Global Impression of Change scale is a single, self-administered question asking respondents to rate how their condition has changed since a certain point in time. It is a patient-reported outcome measure that can be used to assess treatment benefit in clinical trials or practice. It is based on the Clinical Global Impression of Change scale, which is an observer-rated scale of symptom severity and treatment response. The scale ranges from 1 (no change or worse) to 7 (a great deal better).
California Verbal Learning Test (CVLT) Aim 2.1 | Baseline to month 6 visit
  The California Verbal Learning Test - Third Edition (CVLT-III) is a comprehensive assessment of verbal learning and memory. It produces a variety of scores, including:
  d' score A raw score that reflects the difference between the hit rate (signal) and the false positive (FP) rate (noise). The d' score is calculated by subtracting the FP rate from the hit rate, after applying a z-transform to each.
  Total RD A score that can range from +4.0 to -4.0. A high score indicates a high number of hits and a low number of FP errors, while a low score indicates a low number of hits and a high number of FP errors.
  Scaled scores Scores that are adjusted for age and gender using the CVLT-3 standardization sample norms.
  T-scores Scores that are derived from scaled scores and demographic information using look-up tables. T-scores are a comparison of an individual's memory performance to what is expected based on their demographics.
Grey matter volumes of the cingulate cortex and other prefrontal cortex regions Aim 2.2 | Baseline and 6 months
  Change in the structural brain MRI baseline grey matter volumes of the cingulate cortex and other prefrontal cortex regions at 6 months.
  The investigators will use linear mixed effect and coefficient measures, and include sex, age, opioid medications, and duration of CP as confounders and as effect modifiers. Investigators will also estimate linear and non-linear trajectories.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Nwaokobia, Principal Investigator — Evon Medics LLC; Evaristus Nwulia, MD, MHS, Principal Investigator — Evon Medics LLC; Tanya Alim, MD, Principal Investigator — Howard University; Haddi Ogunsola, MD, Principal Investigator — Global Pain Management, LLC
Locations (2):
- United States (2):
  - Howard University, Washington D.C., District of Columbia
  - Global Pain Management LLC, Pasadena, Maryland

IPD SHARING:
Plan to Share IPD: No